CLINICAL TRIAL: NCT03220451
Title: Pilot Study on the Use of Adhesive Elastic Taping as "add-on" Treatment for the Therapy of Medium/Severe Grade Pressure Ulcers in Spinal Cord Injured Patients
Brief Title: Use of Adhesive Elastic Taping for the Therapy of Medium/Severe Pressure Ulcers in Spinal Cord Injured Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montecatone Rehabilitation Institute S.p.A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE-17083
Record Dates: First submitted 2017-07-11; First posted 2017-07-18 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Pressure Ulcer; Spinal Cord Injuries
Keywords: pressure ulcer; pressure sore; decubitus ulcer; spinal cord injury; adhesive elastic bandage; taping; kinesio taping; neuro taping
MeSH Terms: conditions — Pressure Ulcer; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adhesive elastic taping (Experimental): After a 4-week observation of the pressure ulcer under investigation, adhesive elastic tape is applied around it for a 4-week period (the tape is changed twice a week), according to a planned application protocol. The ulcer is then observed for a subsequent follow-up period of 4 weeks.
  Interventions: Procedure: Adhesive elastic taping

INTERVENTIONS:
Procedure: Adhesive elastic taping — Adhesive elastic taping placed around a pressure ulcer, according to a planned placement technique

SUMMARY:
All patients with a significant deficiency of skin sensitivity and reduced mobility are potentially at risk of Pressure Ulcers (PUs), in particular the persons affected by Spinal Cord Injury (SCI), also due to their frequent alteration or loss of subcutaneous skin sensitivity. Pressure sores are one of the most common and fearful complications in SCI, with a severe impact on quality of life and on care health costs. They are often the cause of lengthening the time of hospitalization, slowing down clinical and rehabilitation programs and re-hospitalization.

PUs, when arisen, heal slowly and, despite the protracted conservative medical therapies, sometimes they do not come to complete healing. Sometimes plastic surgery is needed, although even after it recurrence rates remain high.

Further treatments have been proposed in addition to the usual medication, however they are characterized by a certain degree of invasiveness and are often conditioned by the availability of specific and sometimes expensive equipment, as well as by the presence of highly qualified personnel. In general, there is also a lack of good quality clinical trials for assessing their effectiveness and safety and they are often not decisive, especially for severe and recalcitrant ulcers.

Among alternative techniques for the healing of skin ulcers in general, the adhesive elastic bandage, also known as "kinesio taping" and already recognized for the treatment of edema, hematoma and scarring, has been proposed. However, specific protocols and published studies are not available for PUs.

The Montecatone Rehabilitation Institute, that hosts the largest Spinal Unit in Italy, pays great attention to the prevention and treatment of PUs in both acute and chronic patients. The rationale for the taping positioning around PUs investigated in this study is to improve lymphatic drainage and reactivation of the superficial bloodstream by increasing interstitial spaces and reducing skin and subcutaneous compression, notoriously compromised in the areas of onset of pressure sores. The total shortage in the literature and in user manuals of taping protocols for PUs supports this preliminary, exploratory, descriptive and uncontrolled pilot study with the primary aim of verifying the safety of a taping treatment for medium/severe grade PUs, "add-on" to the usual care. The choice of the ulcer sites selected (sacral and heel) has been affected by the feasibility of tape positioning.

DETAILED DESCRIPTION:
All patients with a significant deficiency of skin sensitivity and reduced mobility are potentially at risk of Pressure Ulcers (PUs), in particular the persons affected by Spinal Cord Injury (SCI), also due to their frequent alteration or loss of subcutaneous skin sensitivity. More than one-third of individuals hospitalized in Spinal Units for rehabilitative treatments following a SCI develop PUs during acute hospitalization and it was also estimated that up to 85% of SCI persons develop at least one PU in the course of their lives. Pressure sores are therefore one of the most common and fearful complications in SCI, with a severe impact on quality of life and on care health costs. They are often the cause of lengthening the time of hospitalization, slowing down clinical and rehabilitation programs and re-hospitalization.

PUs, when arisen, heal slowly and, despite the protracted conservative medical therapies, sometimes they do not come to complete healing. Sometimes plastic surgery is needed, although even after it recurrence rates remain high.

Traditional treatment of PUs consists in the use of advanced dressings that may vary depending on the degree of staging of the lesion, its extent and the presence of clinical signs of necrosis and/or deep soft tissue infection. In addition to dressings, treatment cycles with intermittent negative pressure therapy can be indicated and the surgical approach (toilets + plastic reconstruction) could be reserved to chronic lesions with no response to traditional dressings or in the case of underlying osteomyelitis.

Alternative treatments (e.g. electrotherapy, pulsed electromagnetic fields, ultraviolet light, infrared radiation, laser therapy, ultrasound, shock waves) have been proposed in addition to the usual medication, however they are characterized by a certain degree of invasiveness and are often conditioned by the availability of specific and sometimes expensive equipment, as well as by the presence of highly qualified personnel. In general, there is also a lack of good quality clinical trials for assessing the effectiveness and safety of such techniques that are often not decisive for healing, especially for severe and recalcitrant lesions.

Among alternative techniques for the healing of skin ulcers in general, the adhesive elastic bandage, also known as "kinesio taping" or "neuro taping" and already recognized for the treatment of edema, hematoma and scarring, has been proposed. However, specific protocols and published studies are not available for PUs.

The Montecatone Rehabilitation Institute hosts the largest Spinal Unit in Italy as for number of beds and patients admitted. In addition to the intensive rehabilitation of SCI patients, great attention is paid to the prevention and treatment of PUs in both acute and chronic patients, involving physicians, physiotherapists and nurses. Some Physical Therapists of the Hospital are trained and experienced in the use of adhesive elastic bandage for various neuromuscular applications and a physiotherapy/nursing team has conceived, under medical supervision, the taping protocol for the PUs therapy proposed in this study. The rationale for such a taping positioning around PUs is to improve lymphatic drainage and reactivation of the superficial bloodstream by increasing interstitial spaces and reducing skin and subcutaneous compression, notoriously compromised in the areas of onset of pressure sores. Therefore, it is considered that, thanks to the normalization of blood and lymphatic flow, the proposed protocol may have a facilitating action to heal such lesions, especially if they are severe and recalcitrant to normal therapies.

The total shortage in the literature and in user manuals of taping protocols for PUs supports this preliminary, exploratory, descriptive and uncontrolled pilot study with the primary aim of verifying the safety of a taping treatment for medium/severe grade PUs, "add-on" to the usual care. The choice of the ulcer sites selected (sacral and heel) has been affected by the feasibility of tape positioning.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury of any aetiology (traumatic and non-traumatic) and any neurological level, both complete and incomplete, occurred at least 3 months before;
* Pressure ulcer occurred at least 1 month before;
* Pressure ulcer staged III or IV, according to the National Pressure Ulcer Advisory Panel and European Pressure Ulcer Advisory Panel (NPUAP/EPUAP) classification;
* Pressure ulcer located in sacral or heel region;
* Pressure ulcer with cleansed bottom;
* Stable clinical conditions;
* Cognitive integrity and full collaboration of the subject.

Exclusion Criteria:

* Ulcerative skin lesion not due to pressure;
* Pressure ulcer with frank signs of infection or suggestive of underlying osteomyelitis;
* Eczema and/or irritated and/or psoriatic skin around the pressure ulcer;
* Ongoing deep venous thrombosis;
* Known allergy to elastic adhesive tape;
* Ongoing neoplasia;
* Uncompensated diabetes with signs of peripheral vasculopathy;
* Evidence of peripheral polyneuropathy;
* Circulatory problems (e.g. severe lower limb artery disease);
* Significant respiratory problems (e.g. with ongoing assisted ventilation);
* Ongoing sepsis;
* Ongoing severe clinical instability;
* Ongoing oral anticoagulant therapy;
* Ongoing pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Onset of possible adverse events due to the taping treatment | Every day, during the 4-week tape application period
  Visual daily monitoring of possible adverse events, due to the adhesive elastic taping treatment
Onset of possible adverse events due to the adhesive elastic taping treatment | Every day, during the 4-week follow-up after the tape application period
  Visual daily monitoring of possible adverse events, due to the adhesive elastic taping treatment
Onset of possible events hindering the healing of the pressure ulcer under investigation, due to the taping treatment | Every day (during the 4-week tape application period)
  Visual daily monitoring of possible events hindering the healing of the pressure ulcer under investigation, due to the adhesive elastic taping treatment
Onset of possible events hindering the healing of the pressure ulcer under investigation, due to the taping treatment | Every day (during the 4-week follow-up after the tape application period)
  Visual daily monitoring of possible events hindering the healing of the pressure ulcer under investigation, due to the adhesive elastic taping treatment

SECONDARY OUTCOMES:
Evolution of the characteristics of the pressure ulcer under investigation | Baseline (initial visit); once a week during the whole study period (12 weeks)
  Pressure ulcer assessment with Bates-Jensen Wound Assessment Tool (BWAT), once a week
Evolution of the characteristics of the pressure ulcer under investigation | Baseline (initial visit); week 4; week 8; week 12
  Photographic shot of the pressure ulcer
Patient's weight | Baseline (initial visit)
  Patient's weight, in kilograms (kg)
Patient's height | Baseline (initial visit)
  Patient's height, in meters (m)
Patient's Body Mass Index (BMI) | Baseline (initial visit)
  Patient's BMI assessment (as one of the nutritional status indicators): Patient's weight and Patient's height are combined as kg/m^2
Change in patient's blood hemoglobin | Baseline (initial visit); week 4; week 8; week 12
  Dosage of blood hemoglobin (as one of the nutritional status indicators): grams per deciliter
Change in patient's blood number of lymphocytes: | Baseline (initial visit); week 4; week 8; week 12
  Dosage of blood number of lymphocytes (as one of the nutritional status indicators): billions per liter
Change in patient's blood albumin | Baseline (initial visit); week 4; week 8; week 12
  Dosage of blood albumin (as one of the nutritional status indicators): grams per deciliter
Change in patient's blood prealbumin | Baseline (initial visit); week 4; week 8; week 12
  Dosage of blood prealbumin (as one of the nutritional status indicators): milligrams per deciliter
Change in patient's blood total proteins | Baseline (initial visit); week 4; week 8; week 12
  Dosage of blood total proteins (as one of the nutritional status indicators): grams per deciliter
Change in patient's blood transferrin | Baseline (initial visit); week 4; week 8; week 12
  Dosage of blood total transferrin (as one of the nutritional status indicators): milligrams per deciliter
Onset of patient's pain | Baseline (initial visit); twice a day, during the whole study period (12 weeks)
  Pain assessment with Numeric Rating Scale (NRS), twice a day (morning and evening) during the whole study period (12 weeks)
Site of patient's pain (if any) | Baseline (initial visit); twice a day, during the whole study period (12 weeks)
  Description of the site of possibly observed pain, twice a day (morning and evening) during the whole study period (12 weeks)
Change of patient's spasticity | Baseline (initial visit); week 2; week 4; week 6; week 8; week 10; week 12
  Spasticity assessment with the Modified Ashworth Scale (MAS)
Tape employed for taping treatment | End of tape application period (week 8)
  Quantification of total tape employed for the taping application treatment for each pressure ulcer (in meters)
Time-operator employed for taping treatment | End of tape application period (week 8)
  Quantification of total time-operator employed for the taping application treatment for each pressure ulcer (in minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Capirossi, MD Spinal U, Principal Investigator — Montecatone Rehabilitation Institute S.p.A.
Locations (1):
- Montecatone Rehabilitation Institute S.p.A., Imola, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided